CLINICAL TRIAL: NCT06244797
Title: Investigation of the Effects of Y-TZF (Horizontal Platelet-Rich Fibrin) on the Period After Impacted Third Molar Tooth Extraction: Randomized Controlled Clinical Study
Brief Title: Investigation of the Effects of H-PRF on the Period After Impacted Third Molar Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: esengul sen (Other)
Responsible Party: Sponsor-Investigator, esengul sen, Assisstant Prof. DDS, Phd, Head of Oral and Maxillofacial Surgery Department, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-KAEK-146
Record Dates: First submitted 2024-01-11; First posted 2024-02-06 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Impacted Third Molar Tooth
Keywords: Impacted Third Molar Tooth, PRF

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- CONTROL GROUP (Placebo Comparator): Patient group in which no material is placed in the extraction socket after impacted tooth extraction. There will be 25 patients in this group.
  Interventions: Procedure: L-PRF and H-PRF; Procedure: Impacted Tooth Removal
- L-PRF (leukocyte-platelet rich fibrin): (Active Comparator): The patient group in which L-PRF will be placed in the extraction socket after impacted tooth extraction. There will be 25 patients in this group. Device information to be used: Electromag M815P centrifuge device.
  Interventions: Procedure: L-PRF and H-PRF; Procedure: Impacted Tooth Removal
- H-PRF (horizontal-platelet rich fibrin) (Active Comparator): The patient group in which H-PRF will be placed in the extraction socket after impacted tooth extraction. There will be 25 patients in this group. Device information to be used: Electromag M815A2 centrifuge device.
  Interventions: Procedure: L-PRF and H-PRF; Procedure: Impacted Tooth Removal

INTERVENTIONS:
Procedure: L-PRF and H-PRF — Blood (10 ml) will be taken from the patient with the help of an intraket in the arm or hand of appropriate size and size. Then, the blood sample taken will be placed in the PRF device for centrifugation and the sample will be centrifuged. According to the type of PRF, the centrifuge settings will be changed.
Procedure: Impacted Tooth Removal — All patients will be operated on by the same surgeon using the same procedure in order to ensure standardization. Following the administration of 2% articaine with 1:200,000 adrenalin for the inferior alveolar and buccal nerve blocks, a full-thickness mucoperiosteal flap will be raised, and the tooth will be extracted. Following the extraction of the tooth, sterile saline irrigation will be used in the socket, and bleeding control measures will be taken.

SUMMARY:
After wisdom teeth are extracted, the patient may have some complaints in the post-operative period. Pain, swelling and edema are some of them. These inflammatory complications are important for patients and surgeons to reduce the risk of complications and ensure postoperative recovery and develop customized strategy. Many studies have been conducted in the literature to minimize these situations encountered after tooth extraction.

DETAILED DESCRIPTION:
Many studies have been conducted in the literature to minimize these situations encountered after tooth extraction. Various regenerative methods are being developed to reduce these complaints of patients. Regenerative treatments include non-steroidal anti-inflammatory drugs (NSAIDs), laser therapy, steroids, ultrasound, and PRF applications.

PRF(platelet-rich fibrin) application placed in the extraction socket is one of the regenerative methods used to reduce these complaints. PRF has a fibrin structure obtained from natural blood tissue, containing abundant platelets and leukocytes. This fibrin matrix contains various growth factors and cytokines, including growth factor-beta1 (TGF-β1), platelet-derived growth factor (PDGF), vascular endothelial growth factor (VEGF), interleukin (IL), as well as platelets and leukocytes. These factors act directly on promoting the proliferation and differentiation of osteoblasts, endothelial cells, chondrocytes, and various fibroblast sources.

It is known that PRF has a beneficial effect in relieving pain and swelling and reducing the incidence of alveolar osteitis after extraction of an impacted lower third molar. Therefore, it is placed in extraction sockets to try to reduce post-operative complications.

PRF applications are also developing in their own right, and one of them is the H-PRF (horizontal PRF) application. Recently, horizontal centrifugation of PRF has been shown to provide better cell layer separation and minimize cell accumulation that prevents uniform cell layer formation on the distal surfaces of centrifuge tubes.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer ASA I individuals between the ages of 18-40

Exclusion Criteria:

* Those who are pregnant or lactating
* Those receiving anticoagulant or antiplatelet drug therapy
* Those who received radiotherapy to the head and face area
* Those who are allergic to local anesthetics and prescribed medications

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esengül ŞEN, Study Director — Tokat Gaziosmanpasa University
Locations (1):
- Tokat Gaziosmanpaşa Üniversitesi, Tokat Province, Kaleardı Neighbourhood, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Majid OW. Submucosal dexamethasone injection improves quality of life measures after third molar surgery: a comparative study. J Oral Maxillofac Surg. 2011 Sep;69(9):2289-97. doi: 10.1016/j.joms.2011.01.037. Epub 2011 Apr 22. PMID 21514710
- [Background] Landry RG, Turnbull RS, Howley T: Effectiveness of benzydamyne HCl in the treatment of periodontal post- surgical patients. Res Clin Forums. 1988, 10:105-18

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No washout or run-in period was used. After enrollment, no participants were excluded or withdrew prior to randomization; all enrolled participants were assigned to an arm.
Period: Overall Study
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin): | H-PRF (Horizontal-platelet Rich Fibrin)
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin): | H-PRF (Horizontal-platelet Rich Fibrin) | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment, measured in years.
  years | 23.88 (5.01) | 24.28 (5.88) | 24.24 (4.64) | 24.13 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 13 | 49
  Male | 8 | 6 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 25 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Facial Swelling (Sum of 3 Linear Distances, mm)
Description: Swelling was evaluated by measuring three linear facial distances: LC-M (lateral canthus to mandibular angle), T-CL (tragus to labial commissure), and T-P (tragus to soft tissue pogonion). The sum of these distances (in mm) was calculated for each participant preoperatively and on postoperative Days 2 and 7. Mean values are reported. Higher values indicate greater swelling.
  Time Frame:
  Postoperative Day 2 and Day 7
  Unit of Measure:
  Millimeters (mm)
  Measure Type:
  Mean
  Measure of Dispersion/Precision:
  Standard Deviation
Time Frame: Postoperative day 2 and day 7
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin): | H-PRF (Horizontal-platelet Rich Fibrin)
Number analyzed (Participants) | 25 | 25 | 25
Millimeters (mm)
  Day 2 | 122.08 (6.02) | 118.55 (7.22) | 116.90 (6.57)
  Day 7 | 119.68 (5.97) | 115.69 (6.68) | 114.23 (6.59)

2. Primary Outcome: Maximum Interincisal Distance (Mouth Opening, mm)
Description: Trismus was assessed by measuring the maximum interincisal distance (mouth opening) with a calibrated ruler. Measurements were recorded on postoperative Days 2 and 7. Lower values indicate more restricted mouth opening.
Time Frame: postoperative day 2 and day 7
Population: All randomized participants who completed trismus assessments at the specified time points
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin): | H-PRF (Horizontal-platelet Rich Fibrin)
Number analyzed (Participants) | 25 | 25 | 25
Millimeters (mm)
  Day 2 | 28.56 (8.94) | 29.48 (5.69) | 31.20 (6.38)
  Day 7 | 38.96 (5.89) | 39.48 (6.18) | 38.92 (6.10)

3. Secondary Outcome: Soft Tissue Healing (Landry Index, 5-point Scale)
Description: Healing was assessed using the Landry index, a 5-point ordinal scale (1 = very poor, 2 = poor, 3 = fair, 4 = good, 5 = excellent). Assessments were performed on postoperative Days 2 and 7 by a blinded examiner. Higher scores indicate better healing.
Time Frame: Postoperative Day 2 and Day 7
Population: All randomized participants who completed the healing assessment at each time point were analyzed. In the L-PRF arm, one participant's postoperative Day 2 and Day 7 Landry index assessments were not recorded due to a documentation error; therefore, 24 participants were analyzed for this outcome in that arm. No imputation was performed.
  The category 'Very poor' (score = 1) was part of the Landry index but was not observed in any participant on both days.
Measure: Count of Participants; unit: Participants
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin): | H-PRF (Horizontal-platelet Rich Fibrin)
Number analyzed (Participants) | 25 | 24 | 25
Participants
  day 2: Poor | 8 | 3 | 6
  day 2:Fair | 14 | 13 | 9
  day 2: Good | 3 | 8 | 9
  day 2: Excellent | 0 | 0 | 1
  day 7: Poor | 0 | 0 | 0
  day 7: Fair | 6 | 1 | 1
  day7 : Good | 15 | 10 | 10
  day 7:Excellent | 4 | 13 | 14
  day 2 and 7:Very poor | 0 | 0 | 0

4. Secondary Outcome: Postoperative Pain (Visual Analog Scale, 0-10)
Description: The patient's pain assessment will be made with a visual analog scale (VAS). According to this evaluation, a line of a certain length is divided into 10 equal parts. 0 = no pain, 5 = moderate pain, and 10 = unbearable pain. This statement will be reported to the patient verbally, and the patient will be asked to mark the severity of his pain on this note. The patient will be asked to mark the severity of pain on the VAS scale at the 6th hour, 24th hour, 1st day, 2nd day, 3rd day, 4th day, 5th day, 6th day, and 7th day, and how often anti-inflammatory drugs should be used. Higher scores will be assessed as a worse outcome.
Time Frame: 6 hours after surgery and postoperative Days 1 through 7
Population: All randomized participants who completed the pain assessment at each time point were analyzed.
Measure: Median (Full Range); unit: Score on a scale (0-10)
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin): | H-PRF (Horizontal-platelet Rich Fibrin)
Number analyzed (Participants) | 25 | 25 | 25
Score on a scale (0-10)
  6 hours | 6 [1 to 10] | 5 [0 to 10] | 6 [0 to 10]
  Day 1 | 5 [1 to 10] | 4 [0 to 8] | 4 [0 to 9]
  Day 2 | 4 [0 to 10] | 3 [0 to 7] | 3 [0 to 9]
  Day 3 | 3 [0 to 8] | 1 [0 to 5] | 1 [0 to 8]
  Day 4 | 2 [0 to 8] | 1 [0 to 5] | 1 [0 to 8]
  Day 5 | 1 [0 to 6] | 0 [0 to 3] | 0 [0 to 6]
  Day 6 | 1 [0 to 9] | 0 [0 to 4] | 0 [0 to 7]
  Day 7 | 0 [0 to 5] | 0 [0 to 3] | 0 [0 to 7]

5. Secondary Outcome: Oral Health-Related Quality of Life (Majid Questionnaire, Total Score 0-42)
Description: QoL was assessed using the Majid questionnaire (each item 0-3; total range 0-42). Higher scores indicate worse QoL. A total score was calculated only on postoperative Day 4; on Day 7 only subscale scores were analyzed (no total score).
Time Frame: Postoperative Day 4
Population: Total QoL was analyzed on Day 4 only; Day 7 had subscales only.
Measure: Mean (Standard Deviation); unit: Score (0-42)
Groups:
- L-PRF (Leukocyte-platelet Rich Fibrin): The patient group in which L-PRF will be placed in the extraction socket after impacted tooth extraction. There will be 25 patients in this group. Device information to be used: Electromag M815P centrifuge device.
  L-PRF and H-PRF: Blood (10 ml) will be taken from the patient with the help of an intraket in the arm or hand of appropriate size and size. Then, the blood sample taken will be placed in the PRF device for centrifugation and the sample will be centrifuged. According to the type of PRF, the centrifuge settings will be changed.
  Impacted Tooth Removal: All patients will be operated on by the same surgeon using the same procedure in order to ensure standardization. Following the administration of 2% articaine with 1:200,000 adrenalin for the inferior alveolar and buccal nerve blocks, a full-thickness mucoperiosteal flap will be raised, and the tooth will be extracted. Following the extraction of the tooth, sterile saline irrigation will be used in the socket, and bleeding control measures will be taken.
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin) | H-PRF (Horizontal-platelet Rich Fibrin)
Number analyzed (Participants) | 25 | 25 | 25
Score (0-42) | 11.56 (6.92) | 10.67 (5.11) | 12.92 (5.96)

6. Secondary Outcome: Oral Health-Related Quality of Life (Majid Questionnaire Subscales; Days With Symptoms, 0-7)
Description: On postoperative Day 7, Majid questionnaire subscales were recorded as days with symptoms in the past week (possible range 0-7 days for each subscale). Higher values indicate worse QoL. We report median (full range) per arm. No total score was calculated at Day 7.
Time Frame: Postoperative Day 7
Population: No total score was calculated at Day 7.
Measure: Median (Full Range); unit: Days (0-7)
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin) | H-PRF (Horizontal-platelet Rich Fibrin)
Number analyzed (Participants) | 25 | 25 | 25
Days (0-7)
  Day 7-Social Isolation | 1 [0 to 3] | 2 [0 to 7] | 1 [0 to 5]
  Day 7-Speaking | 1 [0 to 7] | 1.5 [0 to 5] | 2 [0 to 4]
  Day 7-Sleeping | 1 [0 to 5] | 1 [0 to 5] | 1 [0 to 4]
  Day 7-Physical appearance | 2 [0 to 7] | 1.5 [0 to 5] | 3 [0 to 5]

7. Secondary Outcome: Oral Health-Related Quality of Life (Majid - Eating & Drinking; Days With Symptoms, 0-7)
Description: On postoperative Day 7, Eating & Drinking difficulty days were recorded (possible range 0-7 days; higher = worse). We report mean ± SD per arm.
Time Frame: Postoperative Day 7
Population: On postoperative Day 7, Eating & Drinking difficulty days were recorded (possible range 0-7 days; higher = worse). We report mean ± SD per arm.
Measure: Mean (Standard Deviation); unit: Days (0-7)
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin) | H-PRF (Horizontal-platelet Rich Fibrin)
Number analyzed (Participants) | 25 | 25 | 25
Days (0-7) | 2.96 (1.49) | 3.17 (2.04) | 3.6 (1.55)

ADVERSE EVENTS:
Time Frame: Postoperative Days 1-7
Description: Adverse events were monitored systematically during the postoperative follow-up period. Patients were asked daily about any unexpected signs or symptoms, and clinical examinations were performed on Days 2 and 7. No definitions differing from ClinicalTrials.gov standards were used.
Arm/Group | CONTROL GROUP | L-PRF (Leukocyte-platelet Rich Fibrin): | H-PRF (Horizontal-platelet Rich Fibrin)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT06244797/Prot_SAP_ICF_000.pdf